CLINICAL TRIAL: NCT03320876
Title: A Multicenter, Open-label, Long-term Extension Safety and Efficacy Study of Filgotinib Treatment in Subjects With Moderately to Severely Active Psoriatic Arthritis.
Brief Title: An Open-label, Long-term Extension Study With Filgotinib in Active Psoriatic Arthritis.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: development program for filgotinib for participants with psoriatic arthritis has been stopped
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-225; 2017-000545-52 (EudraCT Number)
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- filgotinib (Experimental)
  Interventions: Drug: filgotinib

INTERVENTIONS:
Drug: filgotinib — one filgotinib oral tablet once daily.

SUMMARY:
This is a Phase 2, multicenter, open-label, single arm, Long Term Extension (LTE) safety, tolerability and efficacy study of filgotinib in subjects with moderately to severely active PsA. It is estimated that approximately 105 subjects will be rolled-over after they have completed the 16 weeks of double-blind treatment in core study GLPG0634-CL-224. Subjects will be administered filgotinib in this study until filgotinib is registered for PsA or until Week 304, whichever occurs first. The LTE study is concluded with a follow-up visit approximately 4 weeks after the last intake of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are ≥18 years of age, having completed the 16 weeks of treatment in the qualifying core study GLPG0634-CL-224 and who may benefit from filgotinib long-term treatment according to the investigator's judgment.
* Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to continue to use highly effective methods of contraception as described in the protocol.
* Able and willing to sign the informed consent form (ICF), as approved by the Independent Ethics Committee (IEC) and agree to the schedule of assessments.

Exclusion Criteria:

* Subjects who are deemed not to be benefitting from the study drug based upon lack of improvement or worsening of their symptoms. Local guidelines for subject treatment need to be followed.
* Persistent abnormal laboratory values associated with the use of the study drug (including and not limited to hematology, liver and renal function values), according to the investigator's clinical judgment.
* Subjects who discontinued the qualifying core study GLPG0634-CL-224 due to safety or tolerability issues.
* Subjects who require immunization with live/live attenuated vaccine.
* Diagnosis of rheumatic autoimmune disease or inflammatory joint disease other than psoriatic arthritis, except for Sjögren's syndrome.
* Subjects with symptoms suggestive of uncontrolled hypertension, congestive heart failure, uncontrolled diabetes, cerebrovascular accident, myocardial infarction, unstable angina, unstable arrhythmia or any other cardiovascular condition since the inclusion to the GLPG0634- CL-224 study.
* Subjects with symptoms suggestive of gastrointestinal tract ulceration and/or active diverticulitis since the inclusion to the GLPG0634-CL-224 study.
* Subjects with symptoms suggestive of possible lymphoproliferative disease including lymphadenopathy or splenomegaly since the inclusion to the GLPG0634-CL-224 study.
* Subjects with symptoms suggestive of malignancy since the inclusion to the GLPG0634-CL-224 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of subjects with adverse events | Between entry visit and 4 weeks after the last dose.
  To asses safety and tolerability of filgotinib.

SECONDARY OUTCOMES:
Proportion of subjects achieving minimal disease activity (MDA) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on MDA in PsA patients.
Proportion of subjects achieving American College of Rheumatology 20 (ACR20) response | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by ACR20 in PsA patients.
Proportion of subjects achieving ACR50 response | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by ACR50 in PsA patients.
Proportion of subjects achieving ACR70 response | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by ACR70 in PsA patients
Proportion of subjects with Psoriatic Arthritis Disease Activity Score (PASDAS) low disease activity (LDA, i.e. PASDAS ≤ 3.2) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by PASDAS in PsA patients.
Proportion of subjects with PASDAS Very Low Disease Activity (VLDA) (i.e. PASDAS ≤1.9) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by PASDAS in PsA patients.
Percentage of patients subjects with PASDAS LDA (i.e. PASDAS ≤3.2) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by PASDAS in PsA patients.
Percentage of patients subjects with PASDAS VLDA (i.e. PASDAS ≤1.9) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by PASDAS in PsA patients.
Change from core baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by DAPSA in PsA patients.
Proportion of subjects with DAPSA remission/LDA (DAPSA ≤14) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by DAPSA in PsA patients.
Proportion of subjects with DAPSA remission (DAPSA ≤4) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PsA as assessed by DAPSA in PsA patients.
Change from core baseline in Psoriasis Area and Severity Index (PASI) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PASI in PsA patients.
Proportion of subjects with PASI50 | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PASI50 in PsA patients.
Proportion of subjects with PASI75 | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PASI75 in PsA patients.
Proportion of subjects with PASI90 | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PASI90 in PsA patients.
Proportion of subjects with PASI100 | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on PASI100 in PsA patients.
Change from core baseline in Physician's global assessment of psoriasis | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the affect of filgotinib on Physician's global assessment of psoriasis in PsA patients.
Change from core baseline in Patient's Global Assessment of psoriasis | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the affect of filgotinib on patient's global assessment of psoriasis in PsA patients.
Change from core baseline in modified Nail Psoriasis Area and Severity Index (mNAPSI) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on mNAPSI in PsA patients assessment of psoriasis in PsA patients.
Change from core baseline in pruritis numeric rating scale (NRS) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on NRS in PsA patients.
Proportion of subjects achieving a pruritis numeric rating scale (NRS) response(improvement in pruritus NRS score of ≥3) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on NRS in PsA patients.
Change from core baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) enthesitis index | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on SPARCC enthesitis index in PsA patients.
Change from core baseline in Leeds Dactylitis Index (LDI) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on Dactilytis in PsA patients.
Change from core baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on physical function in PsA patients.
Change from baseline in Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-Fatigue scale) | W4, W52, W100, W148, W172, W196, W220, W244, W268, W292, W304.
  To assess the effect of filgotinib on FACIT-Fatigue scale in PsA patients.
Change from core baseline in 36-item Short-Form Health Survey (SF-36) | W4, W52, W100, W148, W172, W196, W220, W244, W268, W292, W304.
  To assess the effect of filgotinib on SF-36 in PsA patients
Change from core baseline in Psoriatic Arthritis Impact of Disease Questionnaire (PsAID). | W4, W52, W100, W148, W172, W196, W220, W244, W268, W292, W304.
  To assess the effect of filgotinib on PsAID in PsA patients.
Change from core baseline in individual components of the ACR response of improvement in multiple disease assessment criteria | At each on-site visit until filgotinib is registered for PsA or until Week 304, whichever occurs first.
  To assess the effect of filgotinib on signs and symptoms of peripheral arthritis and physical function in PsA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Rajendran, MD, Study Director — Galapagos NV
Locations (25):
- ULB Hopital Erasme, Service de Rheumatology, Brussels, Belgium
- Bulgaria (4):
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - UMHAT "SofiaMed", OOD, Block 1, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
- Czechia (2):
  - CCBR Czech, a.s, Pardubice
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Estonia (3):
  - Center for Clinical and Basic Research, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - OÜ Innomedica, Tallinn
- Poland (4):
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól
  - Ai Centrum Medyczne sp. z o.o. sp.k., Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Przychodnia Specjalistyczna, Torun
  - Centrum Medyczne AMED, Warszawa Targowek, Warsaw
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Servicio de Reumatologia, Fuenlabrada
  - Hospital Infanta Luisa, Servicio de Reumatologia, Seville
- Ukraine (9):
  - CI of Healthcare Kharkiv CCH #8 Dept of Rheumatology Kharkiv MA of PGE of MOHU, Ch of Cardiology and Funct Diagnostics, Kharkiv
  - CNI Consultative and Diagnostic Center of Pecherskyi District of Kyiv, Department of Therapy, Kiev
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Unit of Non-coronary HD&Rh, Kyiv
  - CH of State Border Service of Ukraine (Military Base 2522) Dept of Therapy, D.Halytskyi Lviv NMU, Ch of Family Medicine & Dermatology, Venereology, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Rheumatology HSEIU UMSA, Ch of Family Medicine and Therapy, Poltava
  - CI of TRC, Ternopil
  - M.I. Pyrogov VRCH Dept of Rheumatology M.I. Pyrogov VNMU, Ch of IM #1, Vinnytsia
  - MCIC MC LLC Health Clinic, Unit of Cardiology and Rheumatology, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Un of Therapy and CRh Dept of Therapy, Vinnytsia

IPD SHARING:
Plan to Share IPD: No